CLINICAL TRIAL: NCT05540834
Title: A Phase 2 Safety, Dose-finding and Efficacy Study Evaluating Viscoelastic Testing (VET) Guided Tissue Plasminogen Activator (tPA) Treatment in Critically-ill Pro-thrombotic Acute Respiratory Failure
Brief Title: Viscoelastic Testing Guided Tissue Plasminogen Activator Treatment in Acute Respiratory Failure
Acronym: VETtiPAT-ARF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: South West Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Anders Aneman, Professor, South West Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICU001
Record Dates: First submitted 2022-08-22; First posted 2022-09-15 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Acute Respiratory Failure; Hypercoagulability; Fibrinolysis Shutdown
MeSH Terms: conditions — Thrombophilia | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: A two stage study evaluating (1) safety and dose-finding of escalating Actilyse (tPA) doses, followed by (2) a randomised, controlled efficacy study of VET-guided Actilyse treatment + standard care VERSUS standard care alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VET guided tPA administration + standard care (Experimental): Actilyse (tPA) will be administered as a 2-hour bolus then low dose infusion over 24 hours (safety and dose-finding stage) and 72 hours (randomised stage). Regular monitoring of the coagulation status and lysis time using VET will enable increases or decreases/cessation of the dose. Prophylactic low molecular weight heparin will continue throughout.
  Interventions: Drug: Alteplase
- Standard care (No Intervention): Patients will receive standard care for their condition including prophylactic low molecular weight heparin. Coagulation status and lysis time monitoring with VET will occur at the same times as the experimental arm.

INTERVENTIONS:
Drug: Alteplase — The enzyme tissue plasminogen activator that cleaves plasminogen to form plasmin.
  Other Names: Tissue plasminogen activator; tPA; Actilyse; Activase
  Arms: VET guided tPA administration + standard care

SUMMARY:
Patients with coronavirus disease (COVID) and non-COVID acute respiratory failure (ARF) may be at an increased risk of thrombosis due to increased clot formation and decreased clot lysis. This two stage study aims to utilise bedside coagulation technology to detect patients at increased risk and guide tPA treatment to maximise efficacy and safety through a personalised approach.

DETAILED DESCRIPTION:
Acute respiratory failure (ARF) due to COVID is associated with an increased risk of thrombosis causing death. Therapeutic heparin administration was not beneficial in the critically ill.

In non-COVID ARF patients, the presence of multiple pulmonary vessel filling defects associated with the severity of disease and patient outcome, and resolved following the administration of the fibrinolytics, streptokinase and urokinase. An early phase I study reported improved oxygenation in patients with severe ARF following administration of plasminogen activators. The rationale for fibrinolytics in ARF has been published previously and is supported by meta-analysis of preclinical studies.

In both non-COVID and COVID associated ARF, defective fibrinolysis has been demonstrated. Standard coagulation tests cannot identify a hypercoagulable state nor assess fibrinolysis whereas viscoelastic testing (VET), a rapid, point-of-care device commonly used in Intensive Care, is able to detect these disorders. Numerous studies have demonstrated that VET is sufficiently sensitive to detect the coagulopathies associated with ARF, with several parameters associating with disease severity.

The VETtiPAT ARF trial uses VET to identify ARF patients with a procoagulant and hypofibrinolytic phenotype, then to guide tPA (Alteplase) administration thus maximising efficacy and safety through a personalised precision medicine approach.

ELIGIBILITY:
Inclusion Criteria:

1. Acute respiratory failure of primary pulmonary infectious or extrapulmonary infectious aetiology with severity graded by the arterial oxygen partial pressure to inspired fraction of oxygen ratio (P/F) as per the Berlin definition: acute onset of hypoxemia with an arterial partial pressure of oxygen (PaO2) to inspired fraction of oxygen (FiO2) ratio of less than or equal to 300 mmHg with positive end expiratory pressure (PEEP) of 5 cm of water (H2O) or greater
2. Requiring admission to Intensive Care
3. Aged 18 - 75 years of age
4. Procoagulant profile on ClotPro (TradeMark) fibrinogen (FIB)-test +/- extrinsic coagulation pathway (EX)-test - above normal range for amplitude at 10 minutes (A10) and/or maximal clot firmness (MCF) at 30 minutes run time
5. Lysis Time on ClotPro tissue plasminogen activator (TPA)-test ClotPro equal to or greater than 365 seconds

Exclusion Criteria:

1. Platelet count <150 x 109/L or a reduction in platelet count of 50% or more in the last 24 hours
2. Body weight < 60 kg
3. Structural intracranial disease e.g. arterio-venous malformation or aneurysm
4. Previous intracranial haemorrhage
5. Ischaemic stroke within 3 months
6. Traumatic cardiopulmonary resuscitation
7. Hypoxaemia from traumatic lung injury
8. Active or recent bleeding
9. Recent surgery, trauma or invasive procedure
10. Systolic blood pressure (BP) > 180 mm Hg
11. Diastolic BP > 100 mm Hg
12. Pericarditis or pericardial fluid
13. Diabetic retinopathy
14. Currently menstruating
15. Pregnancy - (beta-human chorionic gonadotropin (HCG) to be performed if of child-bearing age)
16. Liver failure (known severe liver disease or an alanine aminotransferase or an aspartate aminotransferase level that is 5 times the upper limit of normal)
17. Kidney failure (estimated Glomerular Filtration Rate (eGFR =<30 mL/hr or receiving renal replacement therapy)
18. Use of therapeutic anticoagulation or platelet antagonists
19. Not for active treatment
20. Unlikely to survive until the day after tomorrow

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in clot lysis time on viscoelastic testing from baseline and up to 72 hours | From start to end of alteplase infusion + 1 and up to 72 hours later/ equivalent timeframe in controls
  The impact of alteplase administration on the clot lysis time (in seconds) measured by the TPA-test using the ClotPro at the bedside

SECONDARY OUTCOMES:
Change in VET coagulation parameters from baseline and up to 72 hours | From start to end of alteplase infusion + 1 and up to 72 hours later/ equivalent timeframe in controls
  The impact of alteplase administration on clot formation related to fibrinogen and the extrinsic pathway (maximum clot firmness (MCF) / amplitude at 10 minutes (A10) in millimeters) measured by the FIB-test and EX-test using the ClotPro at the bedside
Changes in oxygenation | From start to end of alteplase infusion/ equivalent timeframe in controls
  Arterial partial pressure of oxygen to inspired fraction of oxygen (P/F) ratio
Rate of participants with bleeding events | From study entry to Day 5
  Any bleeding events Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or greater
Rate of thromboembolic events | From study entry to Day 30 or hospital discharge, whichever occurs first
  Any thromboembolic event
Changes in organ function | From start to end of alteplase infusion/ equivalent timeframe in controls
  Sequential Organ Failure Assessment (SOFA) score from 0 (normal) to a range of 1-4 with higher scores indicating more severe organ dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Anders Aneman, Principal Investigator — Sydney WAHS
Locations (1):
- Intensive Care Unit, Liverpool Hospital, South Western Sydney Local Health District, Liverpool, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coupland LA, Rabbolini DJ, Schoenecker JG, Crispin PJ, Miller JJ, Ghent T, Medcalf RL, Aneman AE. Point-of-care diagnosis and monitoring of fibrinolysis resistance in the critically ill: results from a feasibility study. Crit Care. 2023 Feb 10;27(1):55. doi: 10.1186/s13054-023-04329-5. PMID 36765421

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT05540834/Prot_SAP_000.pdf